CLINICAL TRIAL: NCT04588818
Title: Adalimumab in Combination With Methotrexate for the Treatment of Non-infectious Panuveitis in Chinese Children
Brief Title: Adalimumab Plus Methotrexate for the Treatment of Pediatric Uveitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, M.D, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-ADA-Uveitis
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Uveitis
Keywords: Pediatric Panuveitis; Methotrexate; Adalimumab
MeSH Terms: conditions — Uveitis | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adalimumab plus Methotrexate (Experimental)
  Interventions: Drug: Adalimumab plus Methotrexate

INTERVENTIONS:
Drug: Adalimumab plus Methotrexate — Adalimumab 40 mg (≥30kg weight) or 20mg (<30kg weight) subcutaneously every other week without loading dose.
  Methotrexate(10 to 20 mg per square meter of body-surface area; maximum dose, 20 mg) .

SUMMARY:
The aim of this study is to determine the efficacy and safety of ADA plus MTX for the treatment in non-infectious pediatric panuveitis.

DETAILED DESCRIPTION:
Although non-infectious uveitis is rare in pediatric population, the irreversible visual impairment due to ocular complications, severe drug adverse effects are disturbing. There is a high rate of chronic disorder of ocular inflammation and unresponsiveness of therapy drugs in pediatric uveitis, which result in structure destruction and functional impairment including band keratopathy, posterior synechiae, cataract, and so on. The systemic and topical glucocorticoid are advocated to control inflammation but carry a high risk of lots of advert events.

Methotrexate is now highly recommended to control uveitis and most commonly prescribed in pediatric uveitis. it was benefit to prolong remission and reduce recurrence. However, despite early intervention 27-48% children do not achieve control of inflammation and 20% experience adverse events. Adalimumab, a fully human anti-tumor necrosis factor α monoclonal antibody, is effective in the treatment of many rheumatic diseases. ADA as the initial treatment in adult patients of uveitis lead to a more optimistic prognosis, a better visual acuity and a lower dose of dosage of daily glucocorticoid.

The investigators propose to test the efficacy and safety of ADA plus MTX for the treatment in non-infectious pediatric panuveitis who were followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-infectious panuveitis
* Age from 2 to 16 years old
* Vision threatening non-infectious uveitis hadn't received standardized systematic treatment before

Exclusion Criteria:

* Patients who had active infection (including hepatitis B or C infection, tuberculosis), malignancy diseases, or bilateral irreversible blindness and any other contraindications of ADA
* previous exposure to another biologic agent

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the time to reach the remission | 12 months

SECONDARY OUTCOMES:
the time of a first relapse once remission | 12 months
macular structure | 12 months
  decrease of central foveal thickness
the total dosage of corticosteriod or the time to steroid discontinuation | 12 months
Best corrected visual Acuityand | 12 months
  increase of BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Teabagy S, Wood E, Bilsbury E, Doherty S, Janardhana P, Lee DJ. Ocular immunosuppressive microenvironment and novel drug delivery for control of uveitis. Adv Drug Deliv Rev. 2023 Jul;198:114869. doi: 10.1016/j.addr.2023.114869. Epub 2023 May 10. PMID 37172782